CLINICAL TRIAL: NCT03070743
Title: Posterior Compression Distraction Reduction Technique System in the Treatment of BI-AAD
Acronym: PCDR-BIAAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Southern Medical University, China (Other)
Responsible Party: Sponsor
Other Study IDs: XW-NS-PCDR
Record Dates: First submitted 2016-10-25; First posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2016-10

CONDITIONS: Basilar Invagination Associated With Atlantoaxial Dislocation
Keywords: basilar invagination; atlantoaxial dislocation; surgery; restoration technique

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PCDR surgery: Posterior Approach Compression Distraction Reduction Surgery is performed.All of patients received this procedure routinely in the department of neurosurgery at Xuanwu Hospital.
  Interventions: Procedure: Posterior Approach Compression Distraction Reduction Surgery

INTERVENTIONS:
Procedure: Posterior Approach Compression Distraction Reduction Surgery — Posterior Approach Compression Distraction Reduction Surgery is performed.All of patients received this procedure routinely in the department of neurosurgery at Xuanwu Hospital.

SUMMARY:
Posterior compression distraction reduction technique （PCDR） in the treatment of Basilar invagination associated with atlantoaxial dislocation

DETAILED DESCRIPTION:
Basilar invagination (BI) refers to the skull base into the direction of cervical spine, mainly to the odontoid process into the foramen magnum is a major change of congenital cranial vertebral junction malformation. Different from trauma or inflammatory lesions, there exists not only in horizontal but also vertical direction dislocation between atlas and axis，At present there is no satisfactory and widely accepted operation method. At present, the main treatment strategy is adopt skull traction to patients preoperative or intraoperative and make vertebra X-ray observation. If the skull traction restored the atlanto-axial dislocation, This case belongs to restorable atlanto-axial dislocation. If the skull traction cannot restore the dislocation, that is non-restorable atlanto-axial dislocation. For the restorable type, posterior occipital cervical internal fixation and fusion should be performed. For the non restorable cases, the main theories is that various ligaments and scars is formed between the anterior arch of atlas and the odontoid process lead to the causes of the longitudinal traction, so transoral anterior atlanto-axial joint lysis is needed first, and then adopt posterior occipital-cervical internal fixation and interbody fusion after the atlanto-axial dislocation is restored. Because the anterior trans-oral atlanto-axial joint lysis has weakness of difficult and high risk, it has limit the popularization of the treatment of atlanto-axial dislocation. Currently only a few several spinal surgery centers have the ability to carry out. Another problem of this treatment strategy is that the function of posterior operation confined to occipital-cervical fixation in situ but not considered the try to adopt the posterior open reduction, this is mainly due to the current clinical application of occipital cervical posterior fixation system be lack of the pressure reduction effect.

Abumi proposed posterior operation incision, atlanto-axial restore intraoperative technique in 1999, and designed the first compression screw that has a restore function in the operation. But it hasn't been widely used because of the intraoperative reposition and internal fixation instrument design is not reasonable and the restore technique has a lot of deficiencies In 2006 Wangchao reported another posterior atlanto-axial dislocation reduction technology. The restore direction of this technology is more reasonable than Abumi's, but the occipital titanium plate adopted in this kind of restore technique is still evolved the occipital-cervical internal fixation system designed by Abumi, just have the mechanical properties of restore level atlanto-axial dislocation. but for atlanto-axial dislocation caused by the Basilar invagination is still need to adopt restore by skull traction. And in many cases also need to perform anterior transoral atlanto-axial joint lysis in order to achieve expected reduction effect.

Wangchao adopt the same occipital-cervical internal fixation system as Abumi technique to perform pressure reduction of atlanto-axial dislocation. This technology is more reasonable in the pressing direction. Using the occipital-cervical internal fixation system was same as Abumi technique it doesn't own the function of Distraction reduction. Therefore for the vertical dislocation of atlanto-axial Still need to restore by skull traction, some patients need the anterior transoral atlanto-axial joint lysis to restore by traction.

In 2010 the members of the project group reported the atlanto-axial dislocation restore by simple posterior screw internal fixation technique and has achieved effect. The investigator can restore vertical dislocation between the atlanto-axial effectively by applying distraction force between occipital screws and axis pedicle screws. For those Basilar Invagination (BI) complicated with Atlanto-axial dislocation(AAD), the rate of Atlanto-axial reduction100% reached 65%. But due to the use of internal fixation system is ordinary occipital cervical internal fixation system （Summit system，DePuy Co) lacking of the function pressure reduction, therefore the effect of level reduction of atlanto-axial dislocation is poor. In some cases it induct atlanto-axial joint rearward opening angle increases, odontoid falling backwards aggregately, the medulla spinal cord angle narrowed further.Furthermore, Part of the reasons why atlanto occipital complex malformation patients failed to achieve 100% reduction is that atlanto-axial lateral is deformities seriously, utual locking, it is difficulty to restore by this technology.

The technology divided intraoperative reduction process into two operating. First of all, restore the level of dislocation between atlanto-axial through pressure, and then restore the vertical dislocation between atlanto-axial through distraction. The investigator designed the compression occipital plate (COP) owned functions both compression and distraction reduction in order to make it convenient in intraoperative technical operation. The investigation report of Patent Bureau indicated that the design of this type of titanium plate is creative and novel.

The clinical application of this technique has achieved initial success in the treatment of basilar invagination complicated with atlanto-axial dislocation patients. This technology so far is the most reasonable posterior reduction technology in the treatment of basilar invagination complicated with atlanto-axial dislocation mechanics mechanism.

Although the compression distraction reduction technology has obvious advantages analyzed from the mechanical properties of angle application of pressurized occipital titanium plate, but if the application of this technology can be safely effective cure basilar invagination and atlanto-axial dislocation patients, improve neurological function, still need further prospective clinical study.

ELIGIBILITY:
Inclusion Criteria:

* CT indicated C0-C1 fusion, ADI>=3mm, CL>=3MM
* Agree with the operation plan
* Agree to be followed up

Exclusion Criteria:

* The pathology is traumatic or RA
* Underwent operations in occipital-cervical region before
* Accompanied with Chiari malformation needed to be decompression
* Perinatal stage
* With mortal diseases
* Without ability to sign papers

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted to the hospital Diagnosed of basilar invagination accompanied with atlantooccipital dislocation.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Storiation of dislocation confirmed by CT and MRI | 1 yr
Firmed bone graft fusion identified by CT | 1 yr
all cause mortality | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Zan Chen, MD, Study Chair — Neurosurgery department, Xuanwu Hospital
Locations (1):
- BEIJING, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided